CLINICAL TRIAL: NCT01730547
Title: Phase 1/2 Clinical Trial With Autologous Mesenchymal Stem Cells for the Therapy of Multiple Sclerosis
Brief Title: Mesenchymal Stem Cells for Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lou Brundin, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSC-MS
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
Keywords: Mesenchymal stem cells; Multiple Sclerosis; Autoimmune diseases
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early treatment with mesenchymal stem cells (Active Comparator): Patients receive a single intravenous dose of autologous bone marrow-derived MSCs followed by placebo at week 24. Fommow up at week 48
  Interventions: Biological: Autologous mesenchymal stem cells
- Delayed treatment with mesenchymal stem cells (Active Comparator): Patients receive placebo for 24 weeks followed by autologous MSCs at week 24, with a follow-up visit at week 48.
  Interventions: Biological: Autologous mesenchymal stem cells

INTERVENTIONS:
Biological: Autologous mesenchymal stem cells

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of autologous mesenchymal stromal cells as treatment for Multiple Sclerosis.

DETAILED DESCRIPTION:
MESEMS is a randomised phase 2 trial done at 15 sites in nine countries. Patients (aged 18-50 years) with active relapsing-remitting or progressive multiple sclerosis were included if they had a disease duration of 2-15 years since onset of multiple sclerosis and an Expanded Disability Status Scale score of 2·5-6·5. Patients were randomly assigned (1:1), according to a crossover design, to receive a single intravenous dose of autologous bone marrow-derived MSCs followed by placebo at week 24, or to receive placebo followed by autologous MSCs at week 24, with a follow-up visit at week 48. Primary objectives were to test safety and activity of MSC treatment. The primary safety endpoint was to assess the number and severity of adverse events within each treatment arm. The primary efficacy endpoint was the number of gadolinium-enhancing lesions (GELs) counted over week 4, 12, and 24 compared between treatment groups. The primary efficacy endpoint was assessed in the full analyis set, after all participants completed the week 24 visit. Efficacy endpoints were evaluated using a predefined statistical testing procedure. Safety was monitored throughout the study by recording vital signs and adverse events at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MS

   a. Relapsing remitting MS (RRMS) not responding to at least a year of attempted therapy with one or more of the approved therapies (beta-interferon, glatiramer acetate, natalizumab, mitoxantrone, fingolimod) as evidenced by one or more of the following: i. ≥1 clinically documented relapse in past 12 months ii. ≥2 clinically documented relapses in last 24 months iii. ≥1 GEL at MRI performed within the last 12 months

   b. Secondary progressive MS (SPMS) not responding to at least a year of attempted therapy with one or more of the approved therapies (beta-interferon, glatiramer acetate, natalizumab, mitoxantrone, fingolimod) as evidenced by both: i. an increase of ≥1 EDSS point (if at randomization EDSS ≤ 5.0) or 0.5 EDSS point (if at randomization EDSS ≥ 5.5) in the last 12 months ii. ≥1 clinically documented relapse or ≥ 1 GEL at MRI within the last twelve months.

   c. Primary progressive MS (PPMS) patients with all the following features: i. an increase of ≥1 EDSS point (if at randomization EDSS ≤ 5.0) or 0.5 EDSS point (if at randomization EDSS ≥5.5), in the last twelve months ii. ≥ 1 GEL at MRI performed within the last 12 months iii. positive cerebrospinal fluid (CSF) (oligoclonal banding)
2. Age 18 to 50 years
3. Disease duration 2 to 10 years (included)
4. EDSS 3.0 to 6.5

Exclusion Criteria:

1. RRMS not fulfilling inclusion criteria
2. SPMS not fulfilling inclusion criteria
3. PPMS not fulfilling inclusion criteria
4. Any active or chronic infection including infection with HIV1-2 or chronic Hepatitis B or Hepatitis C
5. Treatment with any immunosuppressive therapy, including natalizumab and fingolimod, within the 3 months prior to randomization
6. Treatment with interferon-beta or glatiramer acetate within the 30 days prior to randomization
7. Treatment with corticosteroids within the 30 days prior to randomization
8. Relapse occurred during the 60 days prior to randomization
9. Previous history of a malignancy other than basal cell carcinoma of the skin or carcinoma in situ that has been in remission for more than one year
10. Severely limited life expectancy by another co-morbid illness
11. History of previous diagnosis of myelodysplasia or previous hematologic disease or current clinically relevant abnormalities of white blood cell counts
12. Pregnancy or risk or pregnancy (this includes patients that are unwilling to practice active contraception during the duration of the study)
13. eGFR < 60 mL/min/1.73m2 or known renal failure or inability to undergo MRI examination.
14. Inability to give written informed consent in accordance with research ethics board guidelines

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02; Primary Completion 2019-05-09 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
To assess the safety of IV therapy with autologous Mesenchymal Stem Cells (MSCs) in MS patients. | 48 weeks
  The primary objective of the study is to assess the safety of IV therapy with autologous MSCs in MS. Number of participants with adverse events will be documented at week 0,4,8,12,16,20,24,28,32,36,40,44,48 post treatment. Co-primary objective of the study is to evaluate the activity of autologous MSCS in MS patients, in terms of reduction as compared to placebo in the total number of contrast-enhancing lesions (GEL) at MRI acquired on conventional 1,5 T MRI scans over 24 weeks.

SECONDARY OUTCOMES:
To gather preliminary information of the efficacy of the experimental treatment in terms of combined MRI activity and clinical efficacy (incidence of relapses and disability progression). | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institute, Karolinska University Hospital Solna, Stockholm, Sweden

REFERENCES:
- [Derived] Uccelli A, Laroni A, Brundin L, Clanet M, Fernandez O, Nabavi SM, Muraro PA, Oliveri RS, Radue EW, Sellner J, Soelberg Sorensen P, Sormani MP, Wuerfel JT, Battaglia MA, Freedman MS; MESEMS study group. MEsenchymal StEm cells for Multiple Sclerosis (MESEMS): a randomized, double blind, cross-over phase I/II clinical trial with autologous mesenchymal stem cells for the therapy of multiple sclerosis. Trials. 2019 May 9;20(1):263. doi: 10.1186/s13063-019-3346-z. PMID 31072380